CLINICAL TRIAL: NCT01716845
Title: SynapDx Autism Spectrum Disorder Gene Expression Analysis Study
Brief Title: SynapDx Autism Gene Expression Analysis Study
Acronym: SAGA
Status: Completed | Type: Observational
Sponsor: SynapDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 12001
Record Dates: First submitted 2012-10-23; First posted 2012-10-30 (Estimated); Last update posted 2014-12-17 (Estimated); Status verified 2014-12

CONDITIONS: Autism
Keywords: autism; autism spectrum disorders; RNA; gene expression; developmental delay
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Learning Disabilities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Development group 1
- Development group 2
- Development group 3
- Validation group

SUMMARY:
This study will prospectively enroll approximately 660 children, at least 18 months and less than 5 years of age, who have been referred to a pediatric developmental evaluation centers. Enrolled children will have blood drawn for RNA gene expression analysis and undergo a clinical evaluation to determine the presence or absence of a diagnosis of ASD.

The sequential co-primary objectives of this study are:

* To develop an algorithm to classify blood RNA gene expression patterns to maximize agreement between the classification and a clinical assessment of presence or absence of Autism Spectrum Disorders (ASD).
* To prospectively assess the clinical sensitivity and specificity of the blood RNA gene expression classification algorithm (the SDX-002 test) in children referred to a developmental evaluation clinic for a possible developmental disorder.

ELIGIBILITY:
Inclusion Criteria:

1. Referred to a developmental evaluation centers for evaluation of a possible developmental disorder, other than isolated motor problems.
2. Age >= 18 months and < 5 years.
3. Parent/legal guardian has been informed about the study and has signed an informed consent form.

Exclusion Criteria:

1. Prior reliable diagnosis of Autism Spectrum Disorder (i.e. prior evaluation by a multi-disciplinary team has already reliably established Autism Spectrum Disorder diagnosis).
2. Unable or unwilling to complete study procedures

Ages: 18 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 18 months to < 5 years referred to a developmental evaluation centers for evaluation of a possible developmental disorder.
Sampling Method: Probability Sample
Enrollment: 660 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
RNA gene expression in peripheral blood | within 30 days of collection

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States